CLINICAL TRIAL: NCT01102231
Title: Phase II Study of Pemetrexed + Cetuximab + Cisplatin With Concurrent Chemoradiotherapy in Stage III Non-small Cell Lung Cancer (NSCLC)
Brief Title: Chemoradiotherapy in Stage III Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-0803
Record Dates: First submitted 2010-04-10; First posted 2010-04-13 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Stage III Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Cetuximab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Chemoradiotherapy
  Interventions: Drug: Chemotherapy; Drug: ERBITUX; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Chemotherapy — Pemetrexed 500 mg/m², D1 (D1=D22, 4 cycles) Cisplatin 75 mg/m², D1 (D1=D22, 4 cycles)
Drug: ERBITUX — The initial dose of cetuximab (ERBITUX) is 400 mg/m² intravenously administered over 120 minutes, followed by 11 weekly infusions at 250 mg/m² IV over 60 minutes
Radiation: Radiotherapy — 66 Gy (2 Gy by fraction, 5 fractions by week)

SUMMARY:
Radiochemotherapy is a standard for the treatment of unresectable stage III non-small cell lung cancer. The investigators goal is to study the efficacy and the toxicity for a promising association of new agents (cetuximab and pemetrexed) with concurrent radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* non-squamous stage III non-small cell lung cancer
* measurable disease (RECIST 1.1)
* ECOG performance status 0-1
* normal organ and marrow function

Exclusion Criteria:

* prior chest radiation therapy
* history of any cancer other than NSCLC (except non-melanoma skin cancer or carcinoma in situ of the cervix) within the last five years.
* Prior therapy with known specific inhibitors of the EGFR.
* history of severe allergic reaction to prior therapy with monoclonal antibodies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Trédaniel, MD, PhD, Principal Investigator — IFCT, GH Paris Saint-Joseph; Françoise Mornex, MD, PhD, Principal Investigator — IFCT, HCL Lyon-Sud
Locations (38):
- France (38):
  - Clinique de l'Europe, Amiens
  - Centre Hospitalier, Annemasse
  - CHU Besancon - Pneumologie, Besançon
  - Bordeaux - Polyclinique Nord, Bordeaux
  - Caen - Centre François Baclesse, Caen
  - Caen - CHU Côte de Nacre, Caen
  - CH, Chartres
  - CH, Cholet
  - CHU, Clermont-Ferrand
  - CH, Colmar
  - Clinique des Cèdres, Cornebarrieu
  - Dijon - CAC, Dijon
  - CHU Grenoble, Grenoble
  - Institut d'Oncologie Hartmann, Levallois-Perret
  - CHU (Hôpital Calmette) - Pneumologie, Lille
  - CH, Longjumeau
  - Clinique des 4 Pavillons, Lormont
  - Hôpital Louis Pradel, Lyon
  - Hôpital Nord, Marseille
  - Centre Hospitalier, Montélimar
  - CHU, Nancy
  - CH, Nevers
  - Centre Hospitalier, Niort
  - APHP - Hopital Tenon - Pneumologie, Paris
  - Hôpital du Val de Grâce, Paris
  - Hôpital Saint-Joseph, Paris
  - Perpignan - Centre Catalan d'Oncologie, Perpignan
  - HCL - Lyon Sud, Pierre-Bénite
  - CHU, Poitiers
  - Centre Hospitalier, Rambouillet
  - Reims - CHU, Reims
  - Institut Jean Godinot, Reims
  - Centre Frederic Joliot, Rouen
  - Centre Etienne Dolet, Saint-Nazaire
  - Hôpitaux Universitaires - Nouvel Hôpital Civil, Strasbourg
  - Suresnes - Hopital Foch, Suresnes
  - Tours - CHU, Tours
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Tredaniel J, Mornex F, Barillot I, Diaz O, Hennequin C, Le Pechoux C, Lavole A, Giraud P, Souquet PJ, Teixeira L, Vaylet F, Zalcman G, Baudrin L, Morin F, Milleron B. [A phase II study of cetuximab, pemetrexed, cisplatin, and concurrent radiotherapy in patients with locally advanced, unresectable, stage III, non squamous, non-small cell lung cancer (NSCLC)]. Rev Mal Respir. 2011 Jan;28(1):51-7. doi: 10.1016/j.rmr.2010.06.027. Epub 2011 Jan 11. French. PMID 21277474
- See also: IFCT official website — http://www.ifct.fr

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemoradiotherapy + Cetuximab: Chemotherapy + cetuximab + radiotherapy
  Chemotherapy: Pemetrexed 500 mg/m², D1 (D1=D22, 4 cycles) Cisplatin 75 mg/m², D1 (D1=D22, 4 cycles)
  ERBITUX: The initial dose of cetuximab (ERBITUX) is 400 mg/m² intravenously administered over 120 minutes, followed by 11 weekly infusions at 250 mg/m² IV over 60 minutes
  Radiotherapy: 66 Gy (2 Gy by fraction, 5 fractions by week)
Period: Overall Study
Arm/Group | Chemoradiotherapy + Cetuximab
Started | 106
Completed | 91
Not Completed | 15
Not completed — Protocol Violation | 3
Not completed — Lack of Efficacy | 2
Not completed — Death | 2
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Did not received the treatment | 4

BASELINE CHARACTERISTICS:
Groups:
- Chemoradiotherapy + Cetuximab: Chemoradiotherapy
  Chemotherapy: Pemetrexed 500 mg/m², D1 (D1=D22, 4 cycles) Cisplatin 75 mg/m², D1 (D1=D22, 4 cycles)
  ERBITUX: The initial dose of cetuximab (ERBITUX) is 400 mg/m² intravenously administered over 120 minutes, followed by 11 weekly infusions at 250 mg/m² IV over 60 minutes
  Radiotherapy: 66 Gy (2 Gy by fraction, 5 fractions by week)
Arm/Group | Chemoradiotherapy + Cetuximab
Number analyzed (Participants) | 106
Age, Continuous [Median (Full Range); unit: years] | 57.32 [30.6 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 67
Region of Enrollment [Number; unit: participants]
  France | 106
Smoker [Count of Participants; unit: Participants] | 100
Stage [Count of Participants; unit: Participants] — Per the 7th edition of UICC/AJCC staging system. The T staging is determined by the size of primary tumour in long axis, or direct extent of the tumour into adjacent structures such as mediastinum or chest wall. The N classification descibes the degree of spread to regional lymph nodes. This remained unchanged in the 7th edition as the new data showed no change in node staging related survival. The M staging defines the presence of metastases beyond regional lymph nodes.
  Stage IIIA: T1 to T3N2M0 and T4N1M0; Stage IIIB: T1 to T4N3M0, Stage IV: T1 to T4 N1toN3 M1
  Participants
    IIIA | 53
    IIIB | 51
    IV | 2
Histological subtype [Count of Participants; unit: Participants]
  Sarcomatoid | 2
  Adenosquamous | 1
  Adenocarcinoma without bronchoalveolar component | 82
  Non Small Cell | 14
  Neuroendocrine carcinoma | 1
  Non Squamous Non Small Cell | 6
ECOG Performance status [Count of Participants; unit: Participants] — PS0 : fully active, able to carry on all pre-disease performance without restriction PS1 : Restricted in physically strenuous but ambulatory and able to carry out work of a light or sedentary nature, e.g. light house work, office work
  Participants
    PS = 0 | 63
    PS = 1 | 43
Unresectability cause [Count of Participants; unit: Participants]
  Anatomical | 100
  Functional | 6

OUTCOME MEASURES:

1. Primary Outcome: Disease-Control Rate
Description: percentage of patients with disease control (complete response + partial response + stable disease) according to RECIST 1.1 criteria Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for Progressive Disease (at least a 20% increase in the sum of diameters of target lesions).
Time Frame: 16 weeks after inclusion
Population: Eligible population
Measure: Count of Participants; unit: Participants
Arm/Group | Chemoradiotherapy + Cetuximab
Number analyzed (Participants) | 99
Participants | 89
Statistical Analysis 1: Comparison: Chemoradiotherapy + Cetuximab; Test type: Other; Proportion difference = 0.905, 95% CI 2-sided [0.846 to 0.964]

2. Secondary Outcome: 18-month Overall Survival Rate
Description: Percentage of patient alive 18 months after registration
Time Frame: 18 months
Population: Eligible population
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Chemoradiotherapy + Cetuximab
Number analyzed (Participants) | 99
percentage of participant | 42.4 [32.6 to 51.9]

3. Secondary Outcome: Progression Free Survival
Description: Progression-free survival is defined as time between date of inclusion and progression or all-cause death.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 52.3 months (median duration of follow-up)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemoradiotherapy + Cetuximab
Number analyzed (Participants) | 99
Months | 14.4 [11.2 to 18.8]

ADVERSE EVENTS:
Time Frame: Adverse event were collected for a patient from the date of signature of his inform consent form until 30 days after the end of his study treatment. Deaths were collected through study completion.
Arm/Group | Chemoradiotherapy + Cetuximab
All-Cause Mortality (participants affected / at risk) | 51/102
Serious Adverse Events (participants affected / at risk) | 26/102
Other Adverse Events (participants affected / at risk) | 100/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiotherapy + Cetuximab (N=102)
Phlebitis superficial (Vascular disorders) | 1 (1)
Pulmonary embolism (Vascular disorders) | 4 (4)
Hypersensitivity (Immune system disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 7 (7)
Death (General disorders) | 1 (1)
Hyperthermia (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hemoglobin decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Oesophagitis (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (5)
Aphasia (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (3)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Dehydratation (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
device related infection (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiotherapy + Cetuximab (N=102)
Alopecia (General disorders) | 14 (28)
Asthenia (General disorders) | 78 (250)
Chest pain (General disorders) | 19 (47)
Edema limb (General disorders) | 7 (10)
Fever (General disorders) | 14 (23)
Vertigo (General disorders) | 6 (10)
Weight loss (General disorders) | 19 (50)
Hemoglobin decreased (Investigations) | 63 (217)
Neutrophil count decreased (Blood and lymphatic system disorders) | 80 (234)
Platelet count decreased (Blood and lymphatic system disorders) | 62 (178)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (94)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 (28)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 39 (94)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 (16)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Neuropathy (Nervous system disorders) | 7 (8)
Paresthesia (Nervous system disorders) | 7 (12)
Conjunctivitis (Eye disorders) | 9 (13)
Tinnitus (Ear and labyrinth disorders) | 10 (28)
Anorexia (Gastrointestinal disorders) | 45 (106)
Constipation (Gastrointestinal disorders) | 39 (83)
Diarrhea (Gastrointestinal disorders) | 23 (34)
dysgueusia (Gastrointestinal disorders) | 6 (8)
dysphagia (Gastrointestinal disorders) | 65 (181)
Gastralgia (Gastrointestinal disorders) | 8 (12)
Nausea (Gastrointestinal disorders) | 76 (217)
Oral mucosal irritation (Gastrointestinal disorders) | 44 (92)
Pyrosis (Gastrointestinal disorders) | 6 (10)
Vomiting (Gastrointestinal disorders) | 37 (69)
Renal failure (Renal and urinary disorders) | 8 (21)
Acne (Skin and subcutaneous tissue disorders) | 23 (80)
Dermatitis (Skin and subcutaneous tissue disorders) | 27 (58)
Dry skin (Skin and subcutaneous tissue disorders) | 30 (92)
Erythema (Skin and subcutaneous tissue disorders) | 21 (46)
Folliculitis (Skin and subcutaneous tissue disorders) | 36 (124)
Paronychia (Skin and subcutaneous tissue disorders) | 7 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (10)
Rash (Skin and subcutaneous tissue disorders) | 32 (114)
Skin disorder (Skin and subcutaneous tissue disorders) | 16 (46)
Hypokalemia (Metabolism and nutrition disorders) | 7 (14)
Mycosis (Infections and infestations) | 6 (7)

LIMITATIONS AND CAVEATS:
Non randomized study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes